CLINICAL TRIAL: NCT00279474
Title: Evaluation of the Effect of Cognitive Behavior Intervention on Psychological Distress of Cancer Patients and Their Family Members
Brief Title: The Effect of Cognitive Behavior Intervention on Psychological Distress of Cancer Patients and Their Family Members
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1951CTIL
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2005-10

CONDITIONS: Cancer
Keywords: cancer patients; family; cognitive behavior; distress
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Behavioral: cognitive-behavior groups

SUMMARY:
The aim of the study is to evaluate the effect of cognitive behavior group intervention with cancer patients and their family members. Around 80 cancer patients and their family members will participate in group intervention and will be compared with 80 controls.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of cognitive behavior group intervention with cancer patients and their family members. Around 80 cancer patients and their family members will participate in group intervention and will be compared with 80 controls (randomized control study). Brief Symptom Inventory,Fatigue inventory, Mini Sleep Questionnaire and repression-sensitization questionnaire will be answered by the participants pre-, post-intervention and after four months.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking

Exclusion Criteria:

* psychiatric condition

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2004-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Reduction in psychological distress, level of fatigue and sleep problems

CONTACTS AND LOCATIONS:
Overall Officials: Miri Cohen, PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Oncology department, Haifa, Israel